CLINICAL TRIAL: NCT01063556
Title: Pharmacokinetics Study of Donepezil HCl in Subjects Receiving Haemodialysis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E2020-J081-107
Record Dates: First submitted 2010-02-01; First posted 2010-02-05 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2010-11

CONDITIONS: End-Stage Renal Disease
Keywords: end-stage renal disease hemodialysis donepezil hydrochloride pharmacokinetics Cross-Over Study
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Donepezil

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: donepezil HCl
- 2 (Experimental)
  Interventions: Drug: donepezil HCl

INTERVENTIONS:
Drug: donepezil HCl — Subjects will receive donepezil HCL 3 mg without haemodialysis. After an interval of over 15 days, the subjects will receive donepezil 3 mg with haemodialysis.
  Arms: 1
Drug: donepezil HCl — Subjects will receive donepezil HCl 3 mg with haemodialysis. After an interval of over 15 days, the subjects will receive donepezil 3 mg without haemodialysis.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of donepezil HCl 3 mg in subjects with end-state renal disease who were receiving haemodialysis.

DETAILED DESCRIPTION:
This is a randomised, single-center, open-label, single-dose, two-period crossover pharmacokinetics study of donepezil HCl tablets 3 mg in subjects receiving haemodialysis. Subjects will be or will not be receiving haemodialysis. After intervals of over 15 days, the subjects will be receiving the other treatment.

ELIGIBILITY:
Inclusion criteria:

Subjects with end-stage renal disease who were receiving haemodialysis. Subject who are able and willing to give written informed consent.

Exclusion criteria:

Subjects with known hypersensitivity to drugs or foods. Subjects with a corrected QT interval greater than 450 msec at Screening period.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: maximum drug concentration in plasma | 0-48 hours
Pharmacokinetics parameter: maximum drug concentration time in plasma | 0-48 hours
Pharmacokinetics parameter: area under the plasma concentration time curve from Time 0 to 48. | 0-48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hirotake Ishigami, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (1):
- Moriya, Ibaraki, Japan